CLINICAL TRIAL: NCT06040385
Title: Effect of Geometric Modifications of Implant Scan Bodies Compared to Conventional Transfer Techniques on Passivity of Mandibular All on Four Restorations
Brief Title: Effect of Geometric Modifications of Implant Scan Bodies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M0203023RP
Record Dates: First submitted 2023-09-04; First posted 2023-09-15 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2023-09

CONDITIONS: Prosthesis Durability
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Intervention Model Description: For group (I):
  For each patient, two final impressions will be made a) Final impression will be done by conventional one-step impression technique.For the same patient, another final impression using unmodified scan bodies will be done by direct intraoral scan technique.
  For group (II):
  For each patient, two final impressions will be made
  a) Final impression will be done by conventional one-step impression technique.For the same patient another final impression using subtractive modified scan bodies will be done by direct intraoral scan technique.
  Conventional impression for both groups will be poured into stone cast with multiunit abutments analogues, then scanned to be as a reference file for each patient.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- • Group I (control group) (Active Comparator): Final impression will be done by conventional one-step impression technique. For the same patient, another final impression using unmodified scan bodies will be done by direct intraoral scan technique.
  Interventions: Device: Implant supported hybrid prosthesis
- • Group II (Test Group) (Active Comparator): Final impression will be done by conventional one-step impression technique. For the same patient another final impression using subtractive modified scan bodies will be done by direct intraoral scan technique
  Interventions: Device: Implant supported hybrid prosthesis

INTERVENTIONS:
Device: Implant supported hybrid prosthesis — For each patient, implant supported mandibular hybrid prosthesis will be fabricated digitally. Frameworks will be tried in patient's mouth, scanned intraorally by intraoral scanner (IOS).

SUMMARY:
The aim of this clinical study will be the effect of geometric modifications of implant scan bodies compared to conventional transfer techniques on passivity of all on four mandibular restorations

DETAILED DESCRIPTION:
The aim of this study will be the effect of geometric modifications of implant scan bodies compared to conventional transfer techniques on passivity of all on four mandibular restorations.

Evaluation method:

The trueness of the final impression and the passivity of the final prosthesis will be evaluated by two methods:

Invitro evaluation For each patient in every group, the standard tessellation language (STL) files of scanned impressions will be superimposed on the reference file to determine the 3D surface, linear, and angular position analysis.

The STL files for both frameworks will be superimposed on the reference file to determine the passivity.

In vivo (Clinical) evaluation Radiographic evaluation using long cone parallel technique will be done for the framework after 6 month (T6) after one year (T12), and after 18 month (T18) from insertion.

ELIGIBILITY:
Inclusion Criteria:

* 1. All selected patients will have four implants placed in the mandibular interforaminal region according to all -on -four concept.

  2. All selected patients have a healthy mucosa and with no clinical complications.

  3. All patients are cooperative and approve the proposed treatment protocol.

Exclusion Criteria:

* 1. Patients who reject to participate in the study. 2. Patients who need implant placement as a result of previous implant failure.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2025-02-16 (Actual)

PRIMARY OUTCOMES:
passivity of the prosthesis | one year
  Radiographic evaluation using long cone parallel technique will be done for the framework
trueness of final impressions | one year
  For each patient in every group, the standard tessellation language (STL) files of scanned impressions will be superimposed on the reference file to determine the 3D surface, linear, and angular position analysis

SECONDARY OUTCOMES:
patient satisfaction | one year
  patient satisfaction will be evaluated using Visual analogue scale questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University ,Faculty of dentistry, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No